CLINICAL TRIAL: NCT03110653
Title: Remifentanil and Hyperalgesia: Gradual Withdrawal Versus Immediate Discontinuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Dr, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: remi074
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia; Pain
MeSH Terms: conditions — Pain | interventions — Remifentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, the anesthesiologist and an external observer will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil (Active Comparator): Remifentanil TCI: gradual withdrawal: reduction of 30% / 15 mins (2 -> 1.4 -> 1 -> 0.7-> 0.5 -> 0.35 -> 0.25 -> 0 ng/ml)
  Interventions: Drug: Remifentanil
- NaCl 0.9% (Placebo Comparator): Remifentanil abrupt discontinuation / NaCl 0.9% (control group with a reduction of 30% /15 mins) (2 -> 1.4 -> 1 -> 0.7-> 0.5 -> 0.35 -> 0.25 -> 0 ng/ml)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Remifentanil — Remifentanil will be continued postoperatively, while being decreased (gradually by 30% every 15 mins)
  Other Names: ultiva
  Arms: Remifentanil
Drug: NaCl 0.9% — NaCl 0.9% will be administered postoperatively, while being decreased by 30% every 15 mins.
  Other Names: physiological serum
  Arms: NaCl 0.9%

SUMMARY:
Modern anesthesia has made a lot of progress, however, postoperative pain remains one of the major problems associated with patient discomfort, prolonged hospital stay and increased health care costs.

Remifentanil is an ultra-short-acting phenylpiperidine opioid analgesic with high lipid solubility and a rapid onset of effect.

Recently, opioid use has also been associated with postoperative opioid-induced hyperalgesia or acute opioid tolerance. An immediate discontinuation of remifentanil has been associated to increased postoperative pain levels.

We would like to investigate whether a gradual post-operative withdrawal of remifentanil is indeed associated with less immediate pain compared to after an abrupt withdrawal in surgical patients undergoing minor surgery.

DETAILED DESCRIPTION:
Modern anesthesia has made a lot of progress, however, postoperative pain remains one of the major problems associated with patient discomfort, prolonged hospital stay and increased health care costs.

Remifentanil is an ultra-short-acting phenylpiperidine opioid analgesic with high lipid solubility and a rapid onset of effect.

It is rapidly metabolized by non-specific blood and tissue esterases, which also ensures rapid recovery. Remifentanil can be given in high doses and is easily titratable. Due to its rapid elimination, a bridge to post-operative analgesia is a necessity when using this drug.

Recently, opioid use has also been associated with postoperative opioid-induced hyperalgesia or acute opioid tolerance. An immediate discontinuation of remifentanil after digestive surgery has been associated to increased postoperative pain levels.

Studies have been done to investigate this phenomenon. Gradual withdrawal of remifentanil seems to be associated with less pain in a rodent population. (4) A recent study by Norwegian colleagues in a human population evaluating two types of pain stimuli seems to confirm this in healthy volunteers. (5) The investigators would like to investigate whether a gradual post-operative withdrawal of remifentanil is indeed associated with less immediate pain compared to after an abrupt withdrawal in surgical patients undergoing minor surgery.

Methods and materials Sample size The primary outcome of the study is to compare the first post-operative demand of analgesic drugs (mins).

Between both groups, we considered a difference of first demand of post-operative analgesia at 35 minutes or more to be of clinical relevance.

Thus, at a two-sided alpha level of 0.05 and power of 90% (Standard deviation 27), the study needs to be conducted on 26 patients, each group consisting of 13 patients.

As data is always lost, the study will be conducted on 30 patients (15 in each group).

Statistical analysis will be done using Mann-Whitney U test.

Blinding procedure and data collection The study is 'double' blinded. Patients, the anesthesiologist and an external observer will be blinded.

A neutral observer will collect data pre-operatively and post-operatively (first 24 hours post-operation).

Concretely, the observer will pre-operatively collect an informed consent form of the patient and, at the same time, asses the patient's state via QoR-40. Both groups will have a remifentanil infusion upon arrival in the PACU. A nurse, independent to the study, will prepare the adequate post-operative syringe (remifentanil diluted at 20 µg/ml or NaCl 0.9%) and will change the syringe according to pre-operative randomization.

Post-operatively, in the PACU, the quantity of morphine used as well as NRS at several times post-operative will be written down.

Once the patient is at the ward, the observer verifies NRS 24 hours post-operatively and, at the same time, patient comfort at 24 hours post-operative will be evaluated through QoR-40 scores.

Study design Protocol Premedication: each group receives alprazolam (0.5 mg) one hour pre-operatively.

Monitoring In both groups, hemodynamic stability will be evaluated by monitoring ECG, heart rhythm, pulse oximetry and (noninvasive) blood pressure, BIS levels, NMT (TOF ratio).

In case blood pressure drops 20% or more from initial measurement, a bolus of ephedrine will be given in both groups.

The total quantity of each drug used will be written down. All drugs are administered intravenously. Different timings will be written down (induction time, incision time, end of surgery time, extubation time).

Group 1 Induction Remifentanil TCI (Minto model) 5 ng/ml Propofol TCI (Schnider model) closed loop (via Toolbox) adjusted to BIS levels between 40-60 Rocuronium 0.6 mg/kg Maintenance Remifentanil TCI (minto model) 5 ng/ml Propofol TCI (Schnider model) closed loop (via Toolbox) adjusted to BIS levels between 40-60 Upon the incision Acetaminophen 1g Diclofenac 1mg/kg Dexamethasone 10 mg Morphine 0.15 mg/kg Rocuronium 0.3 mg/kg

End of the surgery Ondansetron 4mg Discontinuation of propofol TCI Extubation based on TOFF ratio > 90% Remifentanil TCI 2ng/ml Post-operative analgesia (PACU) Remifentanil TCI: gradual withdrawal: reduction of 30% / 15 mins (2 -> 1.4 -> 1 -> 0.7-> 0.5 -> 0.35 -> 0.25 -> 0 ng/ml) Acetaminophen 1g/6h Diclofenac 1mg/kg /12h Morphine (two mg /5 min if NRS > 3/10) (As all patients are monitored and under immediate medical surveillance, no limit will be imposed to morphine consumption.)

Group 2 Induction Remifentanil TCI (Minto model) 5 ng/ml Propofol TCI (Schnider model) closed loop (via Toolbox) adjusted to BIS levels between 40-60 Rocuronium 0.6 mg/kg Maintenance Remifentanil TCI (Minto model) 5 ng/ml Propofol TCI (Schneider model) closed loop (via Toolbox) adjusted to BIS levels between 40-60 Upon the incision Acetaminophen 1g Diclofenac 1mg/kg Dexamethasone 10 mg Morphine 0.15 mg/kg Rocuronium 0.3 mg/kg

End of the surgery Ondansetron 4mg Discontinuation of propofol TCI Remifentanil TCI 2 ng/ml Extubation based on TOFF ratio > 0.9 Post-operative analgesia (PACU) Remifentanil abrupt discontinuation / NaCl 0.9% (control group with a reduction of 30% /15 mins) (2 -> 1.4 -> 1 -> 0.7-> 0.5 -> 0.35 -> 0.25 -> 0 ng/ml) Acetaminophen 1g/6h Diclofenac 1mg/kg /12h Morphine (two mg / 5 min if NRS > 3/10) (As all patients are monitored and under immediate medical surveillance, no limit will be imposed to morphine consumption.)

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a thyroid surgery
* male/female
* from the age of 18 until 65
* ASA physical status of I-III
* Knowledge of French, English or Dutch is required in order to be enrolled in this study.

Exclusion Criteria:

* Pregnancy
* hypo-/hyperthyroidism
* gastro-duodenal ulcer
* allergy or contraindications to one of the study drugs
* renal insufficiency
* liver insufficiency
* neuropsychiatric disturbance
* BMI >30
* history of drug and alcohol abuse
* preoperative analgesic drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
First demand of postoperative analgesic | 24 hours postoperative
  the first demand of post-operative analgesic will be compared in both groups.

SECONDARY OUTCOMES:
Pain evaluation | 24 hours postoperative
  Numeric Rating Scale (NRS) will be collected multiple times in both groups ( 0,15, 30, 45, 60, 75, 90, 105, 120 minutes, 4 hours and 24 hours postoperatively)
Patient satisfaction | 24 hours postoperative
  A questionnaire (QoR-40) will be given to each patient pre- and post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Barvais, Principal Investigator — Erasme Hospital, Brussels
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saxena S, Gonsette K, Terram W, Huybrechts I, Nahrwold DA, Cappello M, Barvais L, Engelman E. Gradual withdrawal of remifentanil delays initial post-operative analgesic demand after thyroid surgery; double-blinded, randomized controlled trial. BMC Anesthesiol. 2019 Apr 25;19(1):60. doi: 10.1186/s12871-019-0731-9. PMID 31027480